CLINICAL TRIAL: NCT06383442
Title: Effects of Different Types of High Intensity Intermittent Training Combined With Resveratrol Supplementation on Oxidative Stress, Metabolic Adaption and Fat Loss in Aged and Overweight Groups
Brief Title: HIIT on Overweight Middle-aged Adults
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N202103041
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Participants were evenly distributed according to a counterbalanced design and divided into three different groups by the body fat percentage of subjects: 1. L-HIIT group: the long-interval HIIT group (4 × 4 min Exercise/4 min Rest), 2. M-HIIT group: the medium-interval HIIT group (8 × 2 min Exercise /2 min Rest), 3. Control group. Target intensities of each interval bout, exercise and rest (Ex./R.), were 85-90% VO2peak/65-70% VO2peak zones, respectively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- M-HIIT (Experimental)
  Interventions: Other: M-HIIT
- L-HIIT (Experimental)
  Interventions: Other: L-HIIT

INTERVENTIONS:
Other: L-HIIT — the long-interval HIIT group (4 × 4 min Exercise/4 min Rest)
  Arms: L-HIIT
Other: M-HIIT — the medium-interval HIIT group (8 × 2 min Exercise /2 min Rest)
  Arms: M-HIIT

SUMMARY:
36 middle-aged with overweight adults were divided into three groups: 1. L-HIIT group: the long-interval HIIT group (4 × 4 min Exercise/4 min Rest), 2. M-HIIT group: the medium-interval HIIT group (8 × 2 min Exercise/2 min Rest), 3. Control group: no exercise intervention. All groups carried out the training stage for 8 weeks (three sessions per week) and the detraining stage for 4 weeks in order to investigate the effects induced by different HIIT interventions on inflammation, metabolic adaptation, anti-fatigue and exercise performance, and fat loss.

DETAILED DESCRIPTION:
Aging, obesity, have been shown to lead to higher oxidative stress and chronic inflammation. However, high-intensity interval training (HIIT) has anti-inflammatory and anti-obesity benefits. Different training prescriptions may also affect improvements. Therefore, this study will explore the optimal HIIT prescription to improve fat, inflammation, metabolism, and exercise performance in overweight middle-aged and older adults. Thirty-six middle-aged with overweight adults were divided into three groups: 1. L-HIIT group: the long-interval HIIT group (4 × 4 min Exercise/4 min Rest), 2. M-HIIT group: the medium-interval HIIT group (8 × 2 min Exercise/2 min Rest), 3. Control group: no exercise intervention. All groups carried out the training stage for 8 weeks (three sessions per week), then the detraining stage for 4 weeks in order to investigate the effects induced by different HIIT interventions on inflammation, metabolic adaptation, anti-fatigue and exercise performance, and fat loss.

ELIGIBILITY:
Inclusion Criteria:

* Recruit people who are overweight or obese (BMI between 24-35) who are 20-65 years old and have no exercise habits in a sitting lifestyle.

Exclusion Criteria:

* If there are any of the following circumstances, they are not allowed to participate in this research and are included in the listing conditions of this case:

  1. Have smoking and drinking habits.
  2. People who have stroke, type 1 and type 2 diabetes, neuromuscular disease, so that they cannot participate in physical activities.
  3. Chronic obstructive lung disease, asthma, interstitial lung disease or alveolar cyst fibrosis.
  4. Metabolic diseases include thyroid disease, kidney disease (kidney, bladder stones) or liver disease.
  5. Those with arrhythmia, a rhythm regulator, severe cardiovascular disease, peripheral vascular disease or cerebrovascular disease.
  6. People with epilepsy and rheumatoid arthritis.
  7. Those who have implanted artificial joints in the past six months and have had recent surgery.
  8. Migraine, acute thrombosis and hernia.
  9. Those who have engaged in strenuous exercise or have muscle aches within 24 hours before the experiment.
  10. People who feel unwell due to other reasons during the experiment.
  11. People with severe food allergies.
  12. Have hospitalization records within three months.
  13. People with cognitive impairment.
  14. Take any drugs that affect the function of the nervous system.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity Test | Primary Outcomes were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  a graded exercise test (GXT) was performed using a stationary bike ergometer (ergo_bike Premium 8i, Flugplatzstr, Germany) to assess the subject's VO2peak
Aerobic Capacity Test | Primary Outcomes were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  All subjects wore polar heart rate belts (Polar Electro Oy, Kempele, Finland) to monitor maximum heart rate during aerobic capacity testing.
Anti-fatigue performance | Primary Outcomes were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  After a standard warm-up, all subjects were assessed with the classical Wingate (WAnT) on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The average relative mean power parameters were recorded.
skinfold thickness | Primary Outcomes were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  The sum of skinfold thickness at seven sites (triceps, chest, subscapular muscle, upper ilium, abdomen, front thigh, and leg) was measured by using a skinfold caliper (Beta Technology, Santa Cruz, California, USA).
Body composition_body fat | Primary Outcomes were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  The multi-frequency principle was applied to measure body composition by using a bioelectrical impedance analyzer (BIA) on an InBody 570 device (In-body, Seoul, South Korea). To perform the measurements, after the subjects' palms and soles were removed from the sensors, the subjects stood on the footing electrodes and held the sensing handles with two hands. During the measurements, the subjects kept their arms open and left their bodies at an angle of 30° without speaking or moving. The subjects also fasted for at least 8 h before the test. The body fat were meansure

SECONDARY OUTCOMES:
Glucose | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  Safety is assessed function of Glucose (70~100 mg/dL)
Triglycerides | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  Safety is assessed function of blood lipid such as Triglycerides (<150 mg/dL)
low-density lipoprotein (LDL) | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  Safety is assessed function of blood lipid such as LDL (0~140mg/dl)
high-density lipoprotein (HDL) | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  Safety is assessed function of blood lipid such as LDL (0~140mg/dl)
creatine kinase (CK) level | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Assess serum CK(Creatine Kinase, U/L) to monitor physiological fitness. Serum CK (U/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
C-reactive protein (CRP) | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Used commercial kit human CRP (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
tumor necrosis factor (TNF)-R1 | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Used commercial kit human TNF-R1 (R & D SYSTEMS, MN USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
TNF-R2 | were measured before the intervention (at week 0), after eight weeks of HIIT intervention (at week 8), and after the following four weeks of detraining (at week 12).
  At designated time points in the recovery period, blood samples were collected with brachial venous catheters. Used commercial kit human TNF-R1 (R & D SYSTEMS, MN USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan